CLINICAL TRIAL: NCT06424821
Title: A Phase II Clinical Study of Cadonilimab in Combination With Chemotherapy as First-Line Treatment for PD-L1 Negative Advanced Non-Small Cell Lung Cancer
Brief Title: Cadonilimab Plus Chemotherapy as First-line Treatment for PD-L1 Negative NSCLC
Acronym: LungCadX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chunxia Su, Director of Clinical Research Center, Shanghai Pulmonary Hospital, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023LY0204
Record Dates: First submitted 2024-05-12; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: NSCLC
Keywords: PD-L1 negative; PD-1/CTLA-4 bispecific antibody

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trial group (Experimental): Cadonilimab (10 mg/kg, IV, every 3 weeks) plus platinum-based chemotherapy (carboplatin [area under the curve (AUC) 5 mg/mL per min, IV] and paclitaxel [175 mg/m2, IV] for squamous NSCLC, or carboplatin [AUC 5 mg/mL per min, IV] and pemetrexed [500 mg/m2, IV] for non-squamous NSCLC) for up to four cycles, followed by maintenance therapy with cadonilimab for squamous NSCLC, and intravenous cadonilimab plus pemetrexed for non-squamous NSCLC
  Interventions: Drug: Cadonilimab

INTERVENTIONS:
Drug: Cadonilimab — Cadonilimab + chemotherapy
  Other Names: Cadonilimab group

SUMMARY:
The goal of this clinical trial is to investigate the efficacy, safety and tolerability of PD-1/CTLA-4 inhibitor (Cadonilimab) combination with chemotherapy as first-line treatment for PD-L1 negative advanced non small cell lung cancer patients. And also explore the potential biomarkers for predicting the efficacy of PD-1/CTLA-4 inhibitor for advanced non small cell lung cancer.

DETAILED DESCRIPTION:
LungCadX is a multi-center, open-label, single-arm, investigator initiated, phase Ⅱ study. Patients received cadonilimab (10 mg/kg, IV, every 3 weeks) plus platinum-based chemotherapy (carboplatin [area under the curve (AUC) 5 mg/mL per min, IV] and paclitaxel [175 mg/m2, IV] for squamous NSCLC, or carboplatin [AUC 5 mg/mL per min, IV] and pemetrexed [500 mg/m2, IV] for non-squamous NSCLC) for up to four cycles, followed by maintenance therapy with cadonilimab for squamous NSCLC, and intravenous cadonilimab plus pemetrexed for non-squamous NSCLC. The primary endpoint was 12-month PFS rate by investigator assessment per RECIST 1.1. Secondary endpoints included PFS, OS, ORR，DoR，DCR, and the safety. Exploratory objective was to assess blood/tumor/urine/faeces tissue for potential biomarkers study. Adverse events will be monitored throughout the trial and graded according to the CTCAE v5.0.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before implementing any trial-related procedures;
* Aged 18-80 years;
* Expected survival of more than 3 months;
* The investigator confirms the presence of at least one measurable lesion according to RECIST 1.1 criteria;
* Wild-type EGFR/ALK;
* Patients with locally advanced (stage IIIb/IIIc), metastatic, or recurrent (stage IV) NSCLC confirmed by histology or cytology, who are not eligible for curative surgery and cannot undergo definitive radiotherapy/chemotherapy, according to the 8th edition of the TNM staging classification by the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer;
* PD-L1 expression in tumor tissue with Tumor Proportion Score (TPS) < 1%;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* No prior systemic anti-tumor treatment for advanced/metastatic disease; patients who have previously received platinum-based adjuvant chemotherapy/radiotherapy, neoadjuvant chemotherapy/radiotherapy, or curative radiotherapy for advanced disease and experienced disease progression more than 6 months after the last treatment can participate in this study;
* Adequate hematologic function, defined as absolute neutrophil count (ANC) >= 1.5 x 10^9/L, platelet count >= 100 x 10^9/L, hemoglobin >= 90 g/L (without transfusion history within 7 days);
* Adequate liver function, defined as total bilirubin level <= 1.5 times the upper limit of normal (ULN) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels <= 2.5 times ULN in all patients, or <= 5 times ULN in patients with liver metastases;
* Adequate renal function, defined as serum creatinine <= 1.5 times ULN;
* Adequate coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) <= 1.5 times ULN; for subjects receiving anticoagulant therapy, INR/PT should be within the range planned by the anticoagulant;
* Women of childbearing potential must have a negative pregnancy test within 7 days before starting treatment, and must use reliable contraceptive measures (such as intrauterine device, contraceptive pills, and condoms) during the trial and for 30 days after the end of the trial; male subjects of reproductive potential must use condoms for contraception during the trial and for 30 days after the end of the trial;
* Willingness to comply with regular follow-up visits and trial requirements.

Exclusion Criteria:

* Currently participating in interventional clinical research treatment;
* Previously received the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs, or drugs targeting another stimulatory or co-inhibitory T-cell receptor (such as CTLA-4, OX-40, CD137);
* Received traditional Chinese medicine or immunomodulatory drugs (such as thymopeptide, interferon, interleukin, etc.) with anti-tumor indications within 2 weeks prior to the first dose;
* Known allergy to the active ingredient or any excipients of Cadonilimab;
* Active hemoptysis, active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, or peritoneal metastasis requiring clinical intervention;
* Uncontrolled pleural effusion/ascites clinically (patients who do not require drainage of effusion or whose effusion does not increase significantly for 3 days can be included);
* Tumor compression of important organs (such as the esophagus) with accompanying symptoms, compression of the superior vena cava, or invasion of mediastinal large blood vessels, heart, etc.;
* History of severe complications such as severe pulmonary or cardiac disease, with any arterial thrombosis, embolism, or ischemia occurring within 6 months prior to enrollment, such as myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack. History of deep vein thrombosis, pulmonary embolism, or any other serious thrombotic events within 3 months prior to enrollment (thrombotic events related to implanted venous infusion ports or catheters, or superficial vein thrombosis are not considered "serious" thrombotic events);
* History of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vasculitis, or glomerulonephritis related to antiphospholipid syndrome; Patients with stable hypothyroidism on replacement therapy with thyroid hormones are eligible to participate in this study; Patients with controlled type 1 diabetes after receiving a stable insulin treatment regimen are eligible to participate in this study;
* Received systemic corticosteroids (> 10 mg/day of prednisone or equivalent) or other systemic immunosuppressive agents (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] drugs) within 2 weeks prior to randomization; Use of topical, ocular, intra-articular, intranasal, and inhaled corticosteroids is allowed;
* Active systemic infections, including tuberculosis (TB) (clinical diagnosis based on clinical history, physical examination, radiographic findings, and TB testing according to local medical practices), hepatitis B (known positive for hepatitis B surface antigen (HBsAg) with HBV DNA >= 1,000 cps/mL or its lower limit of reference range), hepatitis C, or human immunodeficiency virus (HIV) (positive for HIV antibody);
* Known presence of mental illness or substance abuse that may affect compliance with trial requirements;
* History of conditions, diseases, treatments, or laboratory abnormalities that may interfere with trial results or hinder the subject's full participation in the study, or as determined by the investigator that participation in the study is not in the best interest of the subject.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-09-04 (Estimated); Study Completion 2025-09-04 (Estimated)

PRIMARY OUTCOMES:
1-year Progression-Free Survival (PFS) rate | 1 year
  The 1-year Progression-Free Survival (PFS) rate refers to the proportion of patients who are alive and without disease progression one year after starting treatment.

SECONDARY OUTCOMES:
Progression-free Survival | up to 60 months
  Progression-free survival measures the length of time during and after treatment that a patient lives with the disease without it progressing.
Overall Survival | up to 100 months
  Overall survival measures the length of time from the start of treatment until death from any cause, indicating the effectiveness of the treatment in prolonging patients' lives.
objective response rate | up to 24 months
  Objective response rate represents the proportion of patients showing a predefined level of tumor shrinkage or disappearance in response to treatment.
duration of response | up to 24 months
  Duration of response refers to the length of time during which a patient's tumor remains in remission or shows a positive response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chunxia Su, Phd, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China
Locations (2):
- China (2):
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - NINGBO No.2 Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Public article
Supporting Information: Study Protocol
Time Frame: 2025.6-2026.6
Access Criteria: send request to research team for access to the data